CLINICAL TRIAL: NCT04379999
Title: Impact of Atorvastatin ± Aspirin on Colorectal Biomarkers in Patients With Lynch Syndrome: a Pilot Study
Brief Title: Atorvastatin ± Aspirin in Lynch Syndrome Syndrome
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Prevent Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-1039
Record Dates: First submitted 2020-01-03; First posted 2020-05-08 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Lynch Syndrome
Keywords: HNPCC; MLH1; MSH2; MSH6; PMS2; EPCAM; LYNCH
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — Atorvastatin; Aspirin

STUDY DESIGN:
Intervention Model Description: One group receives atorvastatin 20 mg, and the other group receives atorvastatin 20 mg+ aspirin 325mg
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atorvastatin (Active Comparator): Atorvastatin (LIPITOR) 20 milligram tablet daily for 6 weeks
  Interventions: Drug: Atorvastatin 20mg
- Atorvastatin and Aspirin (Active Comparator): Atorvastatin (LIPITOR) 20 milligram tablet and Aspirin 325 mg tablet daily for 6 weeks
  Interventions: Drug: Atorvastatin 20mg AND Aspirin 325 mg

INTERVENTIONS:
Drug: Atorvastatin 20mg — No history of colorectal cancer and no colorectal adenomas within 5 years.
  Other Names: Lipitor 20mg
  Arms: Atorvastatin
Drug: Atorvastatin 20mg AND Aspirin 325 mg — History of colorectal cancer and/or history of colorectal adenomas within 5 years.
  Other Names: Lipitor 20mg AND Aspirin 325mg
  Arms: Atorvastatin and Aspirin

SUMMARY:
The goal of this study is to investigate that a common cholesterol lowering agent (atorvastatin) alone or combining with a nonsteroidal anti-inflammatory drug (aspirin) would reduce the risk of colorectal cancer (CRC) in high-risk individuals with Lynch syndrome.

DETAILED DESCRIPTION:
This is an exploratory biomarker trial to assess the ability of atorvastatin (common cholesterol lowering agent) alone or combining with aspirin (a nonsteroidal anti-inflammatory drug) to reduce the risk of colorectal cancer in high-risk individuals with Lynch Syndrome. Subjects will be stratified based on their prior history of polyps/cancer to receive atorvastatin without or with aspirin for 6 weeks. Blood and normal colon biopsies will be obtained at Day 0 and at 6 weeks on study. Tissue endpoints for analysis include cell proliferation, apoptosis and changes in gene expression. Circulating lipid profiles and metabolic function, and post-treatment questionnaires will be used to assess the acceptability of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are 18 years of age or older
* Able to read and sign an informed consent document in English
* Eligible subjects will have molecular evidence of Lynch Syndrome (mutation in MLH1, MSH2, MSH6, EPCAM or PMS2)
* History of colorectal cancer if surgically cured and > 1 year from completion of adjuvant chemotherapy

Exclusion Criteria:

* Are <18 years of age
* Unable to read and sign an informed consent document in English
* Have active cancer or are less than 3 years post hormonal maintenance therapy for cancer
* Have statin intolerance or contraindication for aspirin or atorvastatin use
* Are pregnant or are actively breast feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Proliferation (Ki-67) and apoptosis (active caspase 3) by immunohistochemical staining | Changes from baseline to 6 weeks
  Effect of Atorvastatin or/and Aspirin on normal colonic proliferation and apoptosis will be evaluated by comparing of immunohistochemical staining of Ki-67 and active caspase 3 using formalin-fixed paraffin-embedded biopsies collected before and at the 6 weeks of drug treatments. Number of positive cells and total number of evaluated cells will be collected for both assays. Data of cells with positive Ki-67 or active caspase 3 will be expressed as % of positive cells (# positive cells/#total evaluated cells x 100). Statistical analyses will be performed to compare the difference between baseline and 6-weeks data.
Genome-wide expression analyses using RNA-Seq | Changes from baseline to 6 weeks
  Effect of Atorvastatin or/and Aspirin on gene expressions in normal colonic epithelial cells will be analyzed using RNA-Seq. Total RNA will be extracted from frozen biopsies. RNASeq libraries will be generated and sequenced on an Illumina platform and analyzed. Differential expression between samples at baseline and 6-weeks of drug treatment will be assessed for statistical significance. Genes with false discovery rat ≤ 0.05 and a fold-change ≥ 2 will be considered significant.

SECONDARY OUTCOMES:
Rate of adherence of healthy patients with Lynch Syndrome to a 6-week of the treatment regimen (atorvastatin ± aspirin). | 6 weeks
  Medication Adherence to the 6-week course of Atorvastatin or/and Aspirin preventive therapy will be assessed by one question in the follow -up survey which participants complete at the end of the study :"Over 6 weeks of preventive therapy, how many Atorvastatin/Aspirin pills did you forget to take?" In addition, participants will be asked to return medication bottle(s) with or without pills. RA will count pills and record number of missing pills in the system.
Frequency of adverse events among patients administered atorvastatin ± aspirin for 6 weeks | 6 weeks
  The adverse event assessment form is used to collect initial and follow-up information for non-serious and serious adverse events for patients participating in the study. Participants are contacted by RA every two weeks to assess side effects and toxicity. A grading scale from 1 to 5 (1-mild, 2-moderate, 3-severy, 4-life-threatining, 5- death related to AE) and causality (1-unrelated, 2-unlikly, 3-possible, 4-probable, 5-definite, NA- not assessed) are recorded for each adverse event (AE) term. Each AE is reviewed by principal investigator and entered into patient's electronic medical record (EMR)
Acceptability of the pilot study intervention and the willingness of the subject to participate in a similar larger study. | 6 weeks
  Acceptability of the study approach 6 Likert-type items (7 point scale) will assess participants' perceptions of various aspects of the study design as a measure of whether changes need to be made to the study methods or design prior to a larger multi-institutional trial. Participants' scores will be summed and a mean score generated. Mean scores > 4 will be considered in the acceptable range. Our threshold target is 75% of participants with a mean score in the acceptable range.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Hall, MD, MS, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underline the results reported in the article , after de-identification
Time Frame: beginning 9 months and ending 3 years following article publication
Access Criteria: Investigators whose proposed use of data has been approved by a review committee identified for this purpose.Proposals should be directed to Michael.Hall@fccc.edu. To gain access, data requestors will need to sign a data access agreement.